CLINICAL TRIAL: NCT04346329
Title: Immune Monitoring of Prophylactic Effect of Hydroxychloroquine in Healthcare Providers Highly Exposed to SARS-Cov-2
Brief Title: Immune Monitoring of Prophylactic Effect of Hydroxychloroquine in Healthcare Providers Highly Exposed to COVID-19
Acronym: Chloroquine UN
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study did not get financed. Never got started.
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Fundación Salud de los Andes (Other)
Responsible Party: Principal Investigator, Carlos Alberto Parra Lopez, Full Professor, Universidad Nacional de Colombia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNAL-COVID-CP
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: COVID
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Phase III double-blind, randomized, placebo-controlled clinical study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Controlled group with placebo medication similar to hydroxychloroquine (loading dose of 800 mg of hydroxychloroquine the first day followed by 400 mg/week for 90 days)
  Interventions: Drug: Placebo oral tablet
- treated (Experimental): hydroxychloroquine with a loading dose of 800 mg of hydroxychloroquine the first day followed by 400 mg/week for 90 days
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Treated group
  Arms: treated
Drug: Placebo oral tablet — Placebo Group
  Arms: Control

SUMMARY:
This is a PILOT STUDY, a Phase III double-blind, randomized, placebo-controlled clinical study in which we assess the clinical effect of the prophylactic administration of hydroxychloroquine vs. placebo to healthcare workers working at our University Hospital (HUN). Participants in each arm (n = 43) will be administered with a unique loading dose of 800 mg of hydroxychloroquine the first day followed by 400 mg/week for 90 days. The population to be studied (uninfected healthcare personnel) will be highly exposed to SARS-CoV-2 infection. An active search should be made for individuals who become infected while participating in the study, hence, once the informed consent form is signed, the molecular test for the diagnosis of SARS-CoV-2 infection by RT-PCR will be carried out every 4 days in order to determine as closely as possible the moment the participant becomes positive. The results of the diagnostic RT-qPCR tests will be confronted with: (i) the results of immune monitoring of at least 30 immunological parameters in leukocytes and in plasma (levels of selected cytokines and chemokines analyzed by automated flow cytometry software and (ii) the daily recording of data for the presence or absence of signs and symptoms associated with SARS-Cov-2 infection. For the recording of immune monitoring 20mL blood samples will be taken at eight-time points throughout the 90 days of the stud.

DETAILED DESCRIPTION:
The personnel responsible for caring of patients infected by the SARS-CoV-2 virus: doctors, nurses and paramedics working at Intensive Care Units (ICUs)), are at high risk of SARS-CoV-2 infection. Epidemiological figures suggest a high morbidity and mortality of doctors responsible for the care of infected individuals, a factor that darkens further the panorama of the current pandemic. The present proposal has two specific aims: (i) to evaluate whether hydroxychloroquine, used prophylactically at low dose (400mg/week for three months), protect against SARS-CoV-2 infection; and (ii) to examine whether exhaustion and senescence of immune system cells are associated to higher risk of SARS-CoV-2 infection. This is a PILOT STUDY, a Phase III double-blind, randomized, placebo-controlled clinical study in which we assess the clinical effect of the prophylactic administration of hydroxychloroquine vs. placebo to healthcare workers working at our University Hospital (HUN). Participants in each arm (n = 43) will be administered with a unique loading dose of 800 mg of hydroxychloroquine the first day followed by 400 mg/week for 90 days. The population to be studied (uninfected healthcare personnel) will be highly exposed to SARS-CoV-2 infection. Taking into account that around 80% do not express symptoms or that these are mild, an active search should be made for individuals who become infected while participating in the study. For this, once the informed consent form is signed, the molecular test for the diagnosis of SARS-CoV-2 infection by RT-PCR will be carried out every 4 days in order to determine as closely as possible the moment the participant become positive. The results of the diagnostic RT-PCR tests will be confronted with: (i) the results of immune monitoring of at least 30 immunological parameters in leukocytes (number and phenotype of: PMN cells, monocytes, T- and B-lymphocytes and NK-cells) and in plasma (levels of IL-2, IL-6, IL-7, IL-10, GM-CSF, TNF-a, IP-10, MCP-1, MIP-IA, IL-1, CRP, Type IFN-alpha and IFN-betta), analyzed by automated flow cytometry software such as tSNE, SPADE, FlowSOM, among others (see attached file); and (ii) the daily recording of data on the presence or absence of signs and symptoms associated with SARS-Cov-2 infection. For the recording of immune monitoring 20mL blood samples will be taken at eight-time points (day 0) and at 8, 15, 21, 30, 45, 60 and 90 days in order to monitor the baseline of immune functionality throughout the 90 days of the study. In summary, this proposal seeks to identify immunological markers of the immune system important for defense against SARS-CoV-2, that may be useful as prognostic markers for clinical response and treatment of patients with COVID-19, and also, to evaluates whether Hydroxychloroquine, used prophylactically, has a role in protecting against SARS-CoV-2 infection in a group of healthcare workers. If hydroxychloroquine, as we all hope, turns out to be an agent that prevent SARS-Cov-2 infection, a significant group of healthcare workers at HUN at risk of becoming ill during the epidemiological peak (expected May 1st), will be protected thanks to their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Be part of the health personnel (intensivist doctor, hospital doctors, nurses, physical therapists and support staff in the care unit) who will work at the HUN in the period of May 1st, 2020 to August 1, 2020
* Be over 18 years old, exposed to patients with COVID-19. Not having symptoms compatible with an acute respiratory infection for the last 21 days.
* Willingness to donate blood samples and for diagnosis and monitoring of SARS-COV-2 infection throughout the study period.
* Have a Smart Phone in order to facilitate permanent communication with you during the duration of the study.
* Signature of informed consent.

Exclusion Criteria:

* Allergy or hypersensitivity to hydroxychloroquine.
* Contraindications to the use of chloroquine (epilepsy, creatinine clearance <30mL / min).
* Be taking (Abiraterone Acetate, Agalsidase, Conivaptan, Dabrafenib, Dacomitinib, Enzalutamide, Idelalisib), or medications that cannot be discontinued.
* Retinal disease.
* Mifepristone, Mitotane, tiripentol.
* Already established hydroxychloroquine treatment.
* Pregnancy or suspected pregnancy.
* Women in breastfeeding.
* Chronic liver disease (Child-Pugh B or C).
* Kidney disease with a Glomerular Filtration Rate of less than or equal to 30mL / min.
* Cardiac, kidney, liver, ophthalmic, neurological or autoimmune disease previously diagnosed.
* Prolongation of the QT segment in the EKG.
* Previous diagnosis of COVID-19.
* Concomitant taking of medications that prolong the QT segment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Adverse effects | six months after administration of hydroxychloroquine or placebo
  Number of participants with treatment-related adverse events as associated administration of hydroxychloroquine or placebo.

SECONDARY OUTCOMES:
Immune-score | six months after administration of hydroxychloroquine or placebo
  Percentage of expression of immune senescence in cells of the immune system of individuals highly exposed to COVID-19 who receive hydroxychloroquine prophylactically vs. placebo.
COVID-19 prevention | six months after administration of hydroxychloroquine or placebo
  Correlate the immunological profile of highly exposed individuals with SARS-CoV-2 with the clinic of COVID-19.
Clinical response | six months after administration of hydroxychloroquine or placebo
  Determine the clinical outcome in observation timeframe of highly exposed personnel when receiving hydroxychloroquine vs. placebo prophylactically.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Facultad de Medicina - Universidad Nacional de Colombia, Bogota, Cundinamarca
  - Universidad Nacional de Colombia, Bogota, Cundinamarca

IPD SHARING:
Plan to Share IPD: No